CLINICAL TRIAL: NCT07312903
Title: An Open Label, Multicenter Study of DPTX3186 to Evaluate Safety, Tolerability, and Pharmacokinetics in Subjects With Known Wnt Pathway Activated Solid Tumors Where No Other Treatments Exist
Brief Title: DPTX3186 in Wnt Pathway Activated Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dewpoint Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DPTX3186-101
Record Dates: First submitted 2025-12-05; First posted 2025-12-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental)
  Interventions: Drug: DPTX3186

INTERVENTIONS:
Drug: DPTX3186 — Once daily (single dose of study drug in the morning in fasted conditions) for 4 consecutive days (4 days on) and 3 days off in a cycle of 28 days

SUMMARY:
This is a first-in human clinical study of DPTX3186 in subjects with Wnt-pathway activated solid tumors where no other treatments exist. The study will evaluate safety, pharmacokinetics, and initial activity of DPTX3186, as well as explore pharmacodynamic parameters to identify potential biomarkers of efficacy

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor and tumor types known to be Wnt-pathway activated (such as colorectal cancer, gastric cancer, lung cancer, and triple negative breast cancer) and no other approved treatment options available.
* At least one measurable target lesion as defined by RECIST v1.1 on CT, PET/CT, or MRI.
* ECOG performance status of 0 or 1.
* Physiological conditions that may prevent absorption of an oral medication including but not limited to colostomy and ileostomy.
* Age ≥18 years (or ≥ age of majority per local regulation)
* Life expectancy ≥3 months
* Willing and able to comply with protocol requirements

Exclusion Criteria:

* Symptomatic or uncontrolled brain metastasis requiring concurrent treatment,
* Another known malignancy that is progressing or requires active treatment within the last 2 years (except basal cell carcinoma, in situ cervical cancer, etc.).
* Inadequate organ function
* Known hypersensitivity to study drug or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events and serious adverse events. | Up to 36 Months
  1. Outcome Measure: Incidence of Treatment Emergent Adverse-Events Measure Description: Number of subjects with treatment-emergent adverse events (TEAEs) Time Frame: up to 36 months
  2. Outcome Measure: Incidence of Serious Adverse Events Measure Description: Number of subjects with serious adverse events (SAEs) Time Frame: up to 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NEXT San Antonio, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia